CLINICAL TRIAL: NCT03999203
Title: A Cross-sectional Study to Measure Cough in Severe Asthma
Acronym: CISA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Collaborators: King's College London (Other)
Responsible Party: Principal Investigator, Liam Heaney, Professor, Queen's University, Belfast
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: B17/03
Record Dates: First submitted 2018-04-12; First posted 2019-06-26 (Actual); Results first posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-02

CONDITIONS: Asthma; Cough
MeSH Terms: conditions — Asthma; Cough | interventions — Citric Acid; Patient Reported Outcome Measures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A - T2 High Severe Asthmatics (Active Comparator): Severe asthmatic patients with eosinophil count ≥ 0.15x10^9/mL andhigh FeNO levels ≥20 ppb.
  Interventions include 24 hour ambulatory cough monitoring (Leicester Cough Monitor), citric acid cough challenge, fractional exhaled nitric oxide (FeNO) testing, patient reported outcome measures and blood, urine and sputum sampling
  Interventions: Drug: Citric acid; Device: Leicester Cough monitor; Other: fractional exhaled nitric oxide testing (FeNO); Other: Patient reported outcome measures
- B - T2 Low Severe Asthmatics (Active Comparator): Severe asthmatic patients with eosinophil count ≤ 0.15x10^9/mL and low FeNO levels <20 ppb.
  Interventions include 24 hour ambulatory cough monitoring (Leicester Cough Monitor), citric acid cough challenge, fractional exhaled nitric oxide (FeNO) testing, patient reported outcome measures and blood, urine and sputum sampling
  Interventions: Drug: Citric acid; Device: Leicester Cough monitor; Other: fractional exhaled nitric oxide testing (FeNO); Other: Patient reported outcome measures
- C - Mild/Moderate Asthmatics (Active Comparator): mild/moderate severe asthmatics (defined as step 2/3 using the GINA classification of severity) recruited from general respiratory clinics in the Belfast HSC Trust Interventions include 24 hour ambulatory cough monitoring (Leicester Cough Monitor), citric acid cough challenge, fractional exhaled nitric oxide (FeNO) testing, patient reported outcome measures and blood, urine and sputum sampling
  Interventions: Drug: Citric acid; Device: Leicester Cough monitor; Other: fractional exhaled nitric oxide testing (FeNO); Other: Patient reported outcome measures
- D - T2 Intermediate (Active Comparator): Severe asthmatic patients with eosinophil count ≥ 0.15x10^9/mL OR high FeNO levels ≥20 ppb.
  Interventions include 24 hour ambulatory cough monitoring (Leicester Cough Monitor), citric acid cough challenge, fractional exhaled nitric oxide (FeNO) testing, patient reported outcome measures and blood, urine and sputum sampling
  Interventions: Drug: Citric acid; Device: Leicester Cough monitor; Other: fractional exhaled nitric oxide testing (FeNO); Other: Patient reported outcome measures

INTERVENTIONS:
Drug: Citric acid — Citric Acid cough challenge to be administered to assess the cough reflex sensitivity in patients
Device: Leicester Cough monitor — Ambulatory cough monitor to assess cough frequency over a 24 hour period
Other: fractional exhaled nitric oxide testing (FeNO) — Measurement of exhaled nitric oxide to give an indication of airway inflammation
Other: Patient reported outcome measures — A number a patient reported outcome measures will be administered including: Asthma control questionnaire (ACQ-5), mini Asthma Quality of Life Questionnaire (mini AQLQ), Leicester Cough Questionnaire (LCQ), Cough Quality of Life Questionnaire (CQLQ), Cough Hypersensitivity Questionnaire (CHQ) and visual analogue scales for severity og cough (VASc) and Urge to Cough (VASu)

SUMMARY:
This study aims to characterise cough in severe asthma through an observational cross-sectional analysis of patients stratified by inflammatory biomarker profile using a number of subjective and objective cough measurement tools.

DETAILED DESCRIPTION:
This study will use a combination of subjective and objective cough measures to assess the frequency of cough as well as its related morbidity in severe asthmatics. Comparisons will be made between T2-High, T2-Low and T2-intermediate patients defined using a composite biomarker profile (blood eosinophil count and FeNO) to assess the role of cough in each and these results will be compared to the transcriptomic and proteomic measurements in the RASP-UK where the same biomarker profiling is being used to define clinical sub-groups of severe asthma. This study aims to also improve characterisation of the T2-Low population and identify possible mechanisms for the pathophysiology of this group.

60 patients are expected to be recruited to the study. Patients will be provided with an information sheet and have a telephone follow-up after at least 24 hours to ask if they remain interested in participation and if so, they will then be asked back for a baseline visit.

Three groups of severe asthmatics will be recruited (as described in appropriate section) and undergo the following procedures:

* Demographic details, height, weight, spirometry, FeNO and vital signs
* Patient reported outcomes:

  * Asthma Mini-Asthma Quality of Life Questionnaire (mini-AQLQ) - abbreviated version of Juniper AQLQ
  * Asthma Control Questionnaire (ACQ-5 (5 questions);
  * Leicester Cough Questionnaire, the Cough-specific quality-of-life Questionnaire and Cough Hypersensitivity Questionnaire will be used to assess the impact of cough;
  * Visual analogue scales (VAS) for cough (VASc) and urge to cough (VASu) will be used as a measure of cough severity.
* Blood samples - a sample of blood will be taken for whole blood transcriptomic and serum analyses
* Citric acid cough challenge test will be used to measure cough reflex sensitivity in each phenotype.
* Spontaneous sputum sample - if patients produce a sputum sample during spirometry or citric acid challenge, this will be recorded and the sample will be retained for sputum differential cell count and storage of processed soluble components.
* On completing the above procedures, patients will be asked to wear a validated ambulatory cough monitor (Leicester Cough Monitor) for a 24-hour period to assess the frequency of cough and if they agree, will be fully instructed in its use.

Patients will be asked to attend a follow-up visit 2 weeks after baseline. The study procedures will remain the same as visit 1 with the exception of collection of clinical samples.

A mild/moderate population will be recruited and undergo the same procedures as the severe group in a baseline visit. No mild/moderate asthmatics will be asked to attend for a follow-up visit.

ELIGIBILITY:
Inclusion Criteria (Severe Asthmatics):

1. Ability and willingness to comply with the study procedures
2. Age ≥18 to ≤75 years at the time of informed consent
3. Severe asthma (as defined by GINA step 4/5 classification of asthma severity) after a detailed systematic assessment
4. History of asthma treatment with high doses of Inhaled Corticosteroids (≥1000 µg beclomethasone dipropionate daily, or equivalent) and an additional controller
5. Three patient groups with severe asthma will be investigated in the study and will be defined as follows:

   T2-High Severe Asthmatics (Group A)
   * Persistent blood eosinophil count ≥0.3x10^9/mL and
   * Persistent high FeNO levels ≥30 ppb and
   * Adherence to inhaled and oral corticosteroid therapy

   T2-Low Severe Asthmatics (Group B)
   * Persistent blood eosinophil count ≤0.2x10^9/Ml and
   * Persistent low FeNO levels (<30ppb)

   T2 - Intermediate Severe Asthmatics (Group D)
   * Persistent blood eosinophil count ≥ 0.3x10^9/mL OR
   * Persistent FeNO levels ≥ 30 ppb

   As stated above, these measurements are made at each clinic visit as part of routine care and will be available on all subjects prior to Inclusion
6. A chest x-ray or CT scan obtained within 12 months before the time of informed consent and showing no new pathology requiring investigation as a potential cause for their cough

Mild/moderate severe asthmatics (who have received a diagnosis of asthma from a physician and are defined as step 2/3 using the BTS/SIGN classification of severity and ACQ<1.5) aged 18-75 years inclusive will be recruited from general respiratory clinics in the Belfast HSC Trust. Patients must have the ability and willingness to comply with study procedures.

Exclusion Criteria:

1. Baseline FEV1 ≤50% of predicted or ≤ 1.0L
2. Asthma exacerbation within 28 days before the time of informed consent or during screening
3. Major episode of infection requiring any of the following:

   * Admission to hospital for ≥24 hours within the 28 days before the time of informed consent
   * Treatment with intravenous antibiotics within the 28 days before the time of informed consent or during Screening
   * Treatment with oral antibiotics within the 14 days before the time of informed consent or during Screening
4. For adults: Active tuberculosis (TB) requiring treatment within the 12 months before the time of informed consent (patients are also required to have no recurrence of symptoms in the 12 months following completion of TB treatment), or
5. Known history of severe clinically significant immunodeficiency, including, but not limited to, human immunodeficiency virus infection and/or currently receiving or have historically received intravenous Ig for treatment for immunodeficiency Note: Immunodeficiency encompasses a wide spectrum of human conditions and/or diseases. A relative IgG deficiency that is thought, but not proven, to be a feature of severe asthma would not be exclusionary for the study.
6. Diagnosis or history of malignancy, or current investigation for possible malignancy
7. Other clinically significant medical disease that is uncontrolled despite treatment or that is likely, in the opinion of the investigator, to require a change in therapy or affect the ability to participate in the study
8. History of alcohol, drug, or chemical abuse that would impair or risk the patient's full participation in the study, in the opinion of the investigator
9. Current smoker or former smoker with a smoking history of >15 pack-years A current smoker is defined as someone who has smoked one or more cigarettes per day (or marijuana or pipe or cigar) for ≥30 days within the 24 months before the time of informed consent and for whom cotinine testing is positive.

   A former smoker is defined as someone who has smoked one or more cigarettes per day (or marijuana or pipe or cigar) for ≥30 days in his or her lifetime (as long as the 30-day total did not include the 24 months before the time of informed consent) and for whom cotinine testing is negative.

   A pack-year is defined as the average number of packs per day times the number of years of smoking.
10. Initiation of or change in allergen immunotherapy within three months before the time of informed consent
11. Treatment with an investigational agent within 30 days of informed consent or 5 half-lives of the investigational agent, whichever is longer
12. Female patients who are pregnant or lactating

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-10-04 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Liam Heaney, MD, Principal Investigator — Queen's University, Belfast; Lorcan McGarvey, MD, Study Chair — Queen's University, Belfast
Locations (1):
- Queen's University Belfast, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- A - T2 High Severe Asthmatics: Severe asthmatic patients with consistent eosinophil count ≥ 0.15x10^9/mL and consistently high FeNO levels ≥20 ppb.
  Interventions include 24 hour ambulatory cough monitoring (Leicester Cough Monitor), citric acid cough challenge, fractional exhaled nitric oxide (FeNO) testing, patient reported outcome measures and blood, urine and sputum sampling
  Citric acid: Citric Acid cough challenge to be administered to assess the cough reflex sensitivity in patients
  Leicester Cough monitor: Ambulatory cough monitor to assess cough frequency over a 24 hour period
  fractional exhaled nitric oxide testing (FeNO): Measurement of exhaled nitric oxide to give an indication of airway inflammation
  Patient reported outcome measures: A number a patient reported outcome measures will be administered including: Asthma control questionnaire (ACQ-5), mini Asthma Quality of Life Questionnaire (mini AQLQ), Leicester Cough Questionnaire (LCQ), Cough Quality of Life Questionnaire (CQLQ), Cough Hypersensitivity Questionnaire (CHQ) and visual analogue scales for severity og cough (VASc) and Urge to Cough (VASu)
- B - T2 Low Severe Asthmatics: Severe asthmatic patients with consistent eosinophil count ≤ 0.15x10^9/mL and consistently low FeNO levels <20 ppb.
  Interventions include 24 hour ambulatory cough monitoring (Leicester Cough Monitor), citric acid cough challenge, fractional exhaled nitric oxide (FeNO) testing, patient reported outcome measures and blood, urine and sputum sampling
  Citric acid: Citric Acid cough challenge to be administered to assess the cough reflex sensitivity in patients
  Leicester Cough monitor: Ambulatory cough monitor to assess cough frequency over a 24 hour period
  fractional exhaled nitric oxide testing (FeNO): Measurement of exhaled nitric oxide to give an indication of airway inflammation
  Patient reported outcome measures: A number a patient reported outcome measures will be administered including: Asthma control questionnaire (ACQ-5), mini Asthma Quality of Life Questionnaire (mini AQLQ), Leicester Cough Questionnaire (LCQ), Cough Quality of Life Questionnaire (CQLQ), Cough Hypersensitivity Questionnaire (CHQ) and visual analogue scales for severity og cough (VASc) and Urge to Cough (VASu)
- D - T2 Intermediate: Severe asthmatic patients with consistent eosinophil count ≥ 0.15x10^9/mL OR consistently high FeNO levels ≥20 ppb.
  Interventions include 24 hour ambulatory cough monitoring (Leicester Cough Monitor), citric acid cough challenge, fractional exhaled nitric oxide (FeNO) testing, patient reported outcome measures and blood, urine and sputum sampling
  Citric acid: Citric Acid cough challenge to be administered to assess the cough reflex sensitivity in patients
  Leicester Cough monitor: Ambulatory cough monitor to assess cough frequency over a 24 hour period
  fractional exhaled nitric oxide testing (FeNO): Measurement of exhaled nitric oxide to give an indication of airway inflammation
  Patient reported outcome measures: A number a patient reported outcome measures will be administered including: Asthma control questionnaire (ACQ-5), mini Asthma Quality of Life Questionnaire (mini AQLQ), Leicester Cough Questionnaire (LCQ), Cough Quality of Life Questionnaire (CQLQ), Cough Hypersensitivity Questionnaire (CHQ) and visual analogue scales for severity og cough (VASc) and Urge to Cough (VASu)
Period: Overall Study
Arm/Group | A - T2 High Severe Asthmatics | B - T2 Low Severe Asthmatics | C - Mild/Moderate Asthmatics | D - T2 Intermediate
Started | 22 | 6 | 19 | 14
Completed | 22 | 6 | 19 | 14
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A - T2 High Severe Asthmatics | B - T2 Low Severe Asthmatics | C - Mild/Moderate Asthmatics | D - T2 Intermediate | Total
Number analyzed (Participants) | 22 | 6 | 19 | 14 | 61
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Each group was analyzed separately Population: Patient groups analysed seperately This was requested as per comments from review
  years
    Age | 60 [50.3 to 67.5] | 53.5 [46 to 60] | 54 [43 to 63] | 57 [54.8 to 65.3] | 55.5 [53.9 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 3 | 8 | 11 | 37
  Male | 7 | 3 | 11 | 3 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 22 | 6 | 19 | 14 | 61
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 22 | 6 | 19 | 14 | 61
BMI [Median (Inter-Quartile Range); unit: kg/m^2] — Each group was analyzed separately Population: Patient groups analysed seperately
  This was requested as per comments from review
  kg/m^2 | 30.4 [27.1 to 35.1] | 28.4 [26.9 to 37.1] | 26.3 [22.8 to 31.2] | 29.6 [26.6 to 33.2] | 29.0 [27.9 to 30.4]
FEV1 (% predicted) [Median (Inter-Quartile Range); unit: Percentage of predicted] — each group was analyzed separately Population: Patient groups analysed seperately This was requested as per comments from review
  Percentage of predicted | 68.5 [62.8 to 87.3] | 87.0 [78.5 to 90.3] | 95 [83 to 106] | 80 [55.8 to 91] | 83.5 [77.1 to 95.0]

OUTCOME MEASURES:

1. Primary Outcome: Cough Frequency Measurement
Description: Objectively measure cough frequency (measured as hours per hour over a 24 hour monitoring period) in different phenotypes of severe asthma and a mild/moderate control group using a validated ambulatory cough monitor (Leicester Cough Monitor)
Time Frame: Baseline
Measure: Geometric Mean (Standard Deviation); unit: coughs per hour over a 24 hour monitorin
Arm/Group | A - T2 High Severe Asthmatics | B - T2 Low Severe Asthmatics | C - Mild/Moderate Asthmatics | D - T2 Intermediate
Number analyzed (Participants) | 22 | 6 | 19 | 14
coughs per hour over a 24 hour monitorin | 6.6 (2.6) | 2.7 (1.6) | 2.5 (4.1) | 12.7 (2.2)

2. Primary Outcome: Cough Reflex Sensitivity (Citric Acid Cough Challenge)
Description: To objectively measure cough reflex sensitivity in different phenotypes of severe asthma and a mild.moderate control group using citric acid cough challenge testing.
  Patients are asked to inhale increasing concentrations of citric acid solutions and the cough response to each is measured in the 15 seconds following. The final outcome endpoint is described as the concentrations needed to cause 2 coughs (C2)
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: M
Arm/Group | A - T2 High Severe Asthmatics | B - T2 Low Severe Asthmatics | C - Mild/Moderate Asthmatics | D - T2 Intermediate
Number analyzed (Participants) | 22 | 6 | 19 | 14
M | 0.125 [0.03 to 0.38] | 0.25 [0.03 to 2.25] | 0.139 [0.03 to 0.40] | 0.125 [0.05 to 0.25]

3. Secondary Outcome: Asthma Control Questionnaire
Description: Assessment of asthma control using subjective questionnaire (asthma control questionnaire) in different phenotypes of severe asthma. Patient responses graded on likert scale with an average score being calculated. A higher score indicates a worse level of asthma control. Score range 0-6
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: Score
Arm/Group | A - T2 High Severe Asthmatics | B - T2 Low Severe Asthmatics | C - Mild/Moderate Asthmatics | D - T2 Intermediate
Number analyzed (Participants) | 22 | 6 | 19 | 14
Score | 1.9 [1 to 3.1] | 1.9 [0.3 to 2.4] | 0.6 [0 to 1.4] | 1.9 [1 to 3.1]

4. Secondary Outcome: Asthma Quality of Life Questionnaire
Description: Assesment of quality of life in asthma as perceived by the patient using this questionnaire in different phenotypes of severe asthma. Patient responses graded on likert scale with an average score being calculated. A higher score indicates a worse level of asthma related quality of life. Score range 1-7
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: Score
Arm/Group | A - T2 High Severe Asthmatics | B - T2 Low Severe Asthmatics | C - Mild/Moderate Asthmatics | D - T2 Intermediate
Number analyzed (Participants) | 22 | 6 | 19 | 14
Score | 4.5 [2.5 to 5.5] | 4.8 [3.5 to 6.4] | 5.9 [5.3 to 6.6] | 4.7 [2.9 to 5.5]

5. Secondary Outcome: Leceister Cough Questionnaire
Description: Assessment of quality of life in relation to cough in different phenotypes of severe asthma. Patient responses graded on likert scale with an average score being calculated from different symptoms domains wihtin the questionnaire. A lower score indicates a worse level of cough related quality of life. Score range 3-21
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: Score
Arm/Group | A - T2 High Severe Asthmatics | B - T2 Low Severe Asthmatics | C - Mild/Moderate Asthmatics | D - T2 Intermediate
Number analyzed (Participants) | 22 | 6 | 19 | 14
Score | 15.2 [11.1 to 18.5] | 18.7 [14.6 to 19.9] | 20 [17 to 20.5] | 14.2 [9.7 to 17.9]

6. Secondary Outcome: Cough Quality of Life Questionnaire
Description: Assessment of quality of life in relation to cough in different phenotypes of severe asthma. Patient responses graded on likert scale with a total score being calculated. A higher score indicates a worse level of cough related quality of life. Score range 28-112
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: Score
Arm/Group | A - T2 High Severe Asthmatics | B - T2 Low Severe Asthmatics | C - Mild/Moderate Asthmatics | D - T2 Intermediate
Number analyzed (Participants) | 22 | 6 | 19 | 14
Score | 61 [53 to 68.3] | 57 [34.5 to 62.3] | 37 [28 to 62] | 56.5 [46.8 to 73.5]

7. Secondary Outcome: Fractional Exhaled Nitric Oxide (FeNO)
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: Parts per billion (ppb)
Arm/Group | A - T2 High Severe Asthmatics | B - T2 Low Severe Asthmatics | C - Mild/Moderate Asthmatics | D - T2 Intermediate
Number analyzed (Participants) | 22 | 6 | 19 | 14
Parts per billion (ppb) | 47 [25.8 to 83.5] | 9.5 [7.5 to 12] | 19 [13 to 34] | 19 [12 to 24.3]

8. Secondary Outcome: Blood Eosinophil Count
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: cells/ul
Arm/Group | A - T2 High Severe Asthmatics | B - T2 Low Severe Asthmatics | C - Mild/Moderate Asthmatics | D - T2 Intermediate
Number analyzed (Participants) | 22 | 6 | 19 | 14
cells/ul | 420 [270 to 550] | 120 [60 to 130] | 260 [140 to 330] | 190 [110 to 280]

ADVERSE EVENTS:
Time Frame: 1 year, 11 months
Arm/Group | A - T2 High Severe Asthmatics | B - T2 Low Severe Asthmatics | C - Mild/Moderate Asthmatics | D - T2 Intermediate
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/6 | 0/19 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/6 | 0/19 | 0/14
Other Adverse Events (participants affected / at risk) | 0/22 | 0/6 | 0/19 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-12): https://cdn.clinicaltrials.gov/large-docs/03/NCT03999203/Prot_SAP_001.pdf